CLINICAL TRIAL: NCT01853800
Title: Single-dose, Open-label, Randomized, 4-way Crossover Study to Compare 10 mg of an Oral Suspension of Rivaroxaban Under Fasting (2 Different Batches) and 20 mg of an Oral Suspension of Rivaroxaban Under Fed Conditions to 10 mg of an Immediate Release Tablet Under Fasting Conditions in Healthy Subjects
Brief Title: Relative Bioavailability of Oral Suspension of Rivaroxaban Compared to Standard Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16886; 2013-001720-19 (EudraCT Number)
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Biological Availability
Keywords: Relative bioavailability; Rivaroxaban
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rivaroxaban (Treatment A) suspension (BN03501), fasted (Experimental): Subjects received single oral dose of Rivaroxaban suspension 10 mg (Treatment A, Batch number BN03501) under fasting conditions in any intervention period.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Rivaroxaban (Treatment B) suspension (BN03501), fed (Experimental): Subjects received single oral dose of Rivaroxaban suspension 20 mg (Treatment B, Batch number BN03501) under fed conditions in any intervention period.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Rivaroxaban (Treatment C) suspension (BR05701), fasted (Experimental): Subjects received single oral dose of Rivaroxaban suspension 10 mg (Treatment C, Batch number BR05701) under fasting conditions in any intervention period.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Rivaroxaban (Treatment D) IR tablet, fasted (Experimental): Subjects received single oral dose of Rivaroxaban IR tablet 10 mg (Treatment D) under fasting conditions in any intervention period.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939)

SUMMARY:
Rivaroxaban is a substance developed for use in the treatment of blood coagulation disorders. Thrombosis (blood clots) can occur as a result of excessive coagulation activity in the blood vessels. Excessive coagulation activity can occur in children as well, and rivaroxaban is therefore being developed for the treatment of thromboembolic events in children and adolescents. As small children are often unable to swallow tablets, an oral suspension (mixture of a liquid containing finely distributed solids) has been developed which allows dosing according to body weight. The objective of this trial is to compare the bioavailability (proportion of a substance that remains available unchanged in the blood circulation) of a rivaroxaban oral solution with that of the rivaroxaban tablet approved for treatment. In order to evaluate the potential influence of food, the oral suspension containing 20 mg rivaroxaban will be taken after consuming food. In addition, the pharmacokinetics (concentrations of the drug and breakdown products (metabolites) in blood), safety and tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age: 18 to 55 years (inclusive) at the first screening examination

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known coagulation disorders (eg von Willebrand's disease, hemophilia)
* Known disorders with increased bleeding risk (eg periodontosis, hemorrhoids, acute gastritis, peptic ulcer)
* Known sensitivity to common causes of bleeding (eg nasal)
* Regular use of medicines
* Clinically relevant findings in the ECG (electrocardiogram) such as a second- or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QTc-interval over 450 msec
* Clinically relevant findings in the physical examination
* Clinically relevant deviations of the screened laboratory parameters from reference ranges
* Participation in another clinical study during the preceding 3 months (Last Treatment from previous study to First Treatment of new study)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Zero to Infinity After a Single Dose (AUC) | 0-72 hours
Area Under the Concentration Versus Time Curve From Zero to Infinity Divided by Dose (AUC/D) | 0-72 hours
Maximum Observed Drug Concentration in Measured Matrix After a Single Dose (Cmax) | 0-72 hours
Maximum Observed Drug Concentration in Measured Matrix Divided by Dose (Cmax/D) | 0-72 hours

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Zero to Infinity Divided by Dose per Kilogram Body Weight (AUC,norm) | 0-72 hours
Area Under the Concentration Versus Time Curve From Zero to Last Quantifiable Concentration [AUC(0tlast)] | 0-72 hours
Maximum Observed Drug Concentration Divided by Dose per Kilogram Body Weight (Cmax,norm) | 0-72 hours
Mean Residence Time (MRT) | 0-72 hours
Maximum Observed Drug Concentration Divided by Drug Concentration at 24 hours (Cmax/C24h) | 0-72 hours
Time to Reach Maximum Observed Drug Concentration (tmax) | 0-72 hours
Terminal Half Life (t1/2) | 0-72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Wuppertal, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/